CLINICAL TRIAL: NCT02722421
Title: A Pharmacokinetic Evaluation of Increased Dose Levonorgestrel Implant and Efavirenz-Based Antiretroviral Therapy In HIV-Infected Ugandan Women
Brief Title: Pharmacologic Strategies to Use the Levonorgestrel Implant in HIV-infected Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Infectious Diseases Institute, Uganda (Other); University of Liverpool (Other); Northwestern University Feinberg School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0234-16-FB; 1R01HD085887-01A1 (NIH)
Record Dates: First submitted 2016-03-02; First posted 2016-03-30 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: HIV; Contraception
Keywords: efavirenz; levonorgestrel; contraceptive implant
MeSH Terms: interventions — Levonorgestrel; efavirenz; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Efavirenz group (Experimental): HIV-infected women receiving efavirenz-based antiretroviral therapy plus increased dose levonorgestrel subdermal implants.
  Interventions: Drug: Levonorgestrel; Drug: Efavirenz

INTERVENTIONS:
Drug: Levonorgestrel — Increased dose levonorgestrel implant plus efavirenz-based antiretroviral therapy.
  Other Names: Jadelle; SinoImplant
Drug: Efavirenz — Participants will receive efavirenz-based ART as part of standard of care
  Other Names: Sustiva; Stocrin; Atripla; EFV

SUMMARY:
The purpose of this study is to determine whether increasing the dose of the levonorgestrel subdermal contraceptive implant will overcome a detrimental drug-drug interaction with efavirenz based antiretroviral therapy.

DETAILED DESCRIPTION:
The investigators research team recently demonstrated that combined use of efavirenz (EFV) based antiretroviral therapy (ART), the only preferred first-line ART regimen in low and middle income countries, with a levonorgestrel (LNG)-releasing implant for one year reduced LNG plasma concentrations by approximately 50% compared to women not on ART. Importantly, the investigators also observed three unintended pregnancies (15%) in the investigators study group of women on EFV-based ART plus the LNG implant, in contrast to the <1% expected failure rate of the implant for women without drug interactions.

This study will determine if increasing the dose of the LNG-releasing subdermal implant effectively overcomes the known pharmacokinetic interaction with EFV- based ART. LNG pharmacokinetic results from the participants enrolled in this dose escalation study (n=28) will be compared to HIV-infected Ugandan women on standard dose LNG without concomitant EFV-based ART.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
2. Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Women age 18 years to 45 years
4. Diagnosed with HIV infection
5. Desiring LNG subdermal implant as a contraceptive method
6. Receiving EFV-based ART for a minimum of 3 months prior to screening
7. Must agree to have concurrent highly effective non-hormonal contraception with a copper intrauterine device (IUD), if not previously medically sterilized.
8. Participants must have a negative urine pregnancy test at entry and report no unprotected sex since the last menstrual period or in the last two weeks.

Exclusion Criteria:

1. HIV RNA > 50 copies/mL at screening visit
2. Serum hemoglobin < 10.0 g/dl
3. Elevations in serum levels of alanine transaminase (ALT) above 5 times the upper limit of normal
4. Elevations in serum creatinine above 2.5 times the upper limit of normal
5. Use of drugs known to be contraindicated with LNG or EFV within 30 days of study entry. Due to the dynamic nature of drug interactions related to ART, the study team will review all concomitant medications at screening based on the US Department of Health and Human Services drug interaction table.
6. Currently pregnant or postpartum <30 days at study entry
7. Concurrent use of other hormonal contraception (Note: use of other forms of hormonal contraception is permissible until time of study enrollment/insertion of LNG implant. Transition from other forms of hormonal contraception to LNG subdermal implant will be accommodated according to LNG product labeling)
8. For the EFV group, participants determined to be ineligible for IUD placement by the World Health Organization (WHO) Medical Eligibility Criteria for Contraceptive Use
9. If participation in the study puts the participant at unacceptable risk based on the judgment of the study staff

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Levonorgestrel plasma concentrations | 24-weeks after implant placement
  We will compare levonorgestrel plasma concentrations between the participants who are receiving increased dose levonorgestrel implants plus efavirenz to historical control participants of HIV-infected Ugandan women not receiving efavirenz.

SECONDARY OUTCOMES:
Levonorgestrel plasma concentrations | 48 weeks after implant placement
  We will compare levonorgestrel plasma concentrations between the participants who are receiving increased dose levonorgestrel implants plus efavirenz to historical control participants of HIV-infected Ugandan women not receiving efavirenz.
Levonorgestrel plasma concentrations | Years 2-3 after implant placement
  This arm will only be continued if safety measures are met at weeks 24 and 48.
Number of adverse events reported by the participant or provider during the study period | 48 weeks after implant placement
  Adverse events reported by participants

OTHER OUTCOMES:
Difference in levonorgestrel concentrations between patients based on pharmacogenetic polymorphisms | 48 weeks after implant placement
  Levonorgestrel PK described by pharmacogenetic polymorphisms
Influence of patient weight (in kg) on levonorgestrel concentrations | 48 weeks after implant placement
  Levonorgestrel PK described by weight
Participant satisfaction with the contraceptive implant reported as a likert scale based on a patient questionnaire | 48 weeks after implant placement
  Patient reported satisfaction with contraceptive method

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly K Scarsi, PharmD, Principal Investigator — University of Nebraska
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No